CLINICAL TRIAL: NCT06697262
Title: Impact of a Telemonitoring Device on the Occurrence of Fever at Home in Children at Risk of Chemotherapy-Induced Neutropenia: A Pilot Randomized Controlled Trial
Brief Title: Impact of a Telemonitoring Device on the Occurever at Home in Children at Risk of Chemotherapy-Induced Neutropenia
Acronym: TELEDOM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024/CHU/03
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Oncopediatrics; Febrile Neutropenia
MeSH Terms: conditions — Febrile Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remote temperature monitoring device (Experimental)
  Interventions: Device: Remote temperature monitoring device
- home temperature monitoring by a nurse (Active Comparator)
  Interventions: Diagnostic Test: Home temperature monitoring by a nurse

INTERVENTIONS:
Device: Remote temperature monitoring device — * Use of the Tucky® remote monitoring device for continuous temperature monitoring at home,
  * In combination with education sessions on temperature monitoring and the device.
  Arms: remote temperature monitoring device
Diagnostic Test: Home temperature monitoring by a nurse — * Home temperature monitoring by a nyrse, twice a day,
  * In association with education sessions on temperature monitoring.
  Arms: home temperature monitoring by a nurse

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility of the study, measured by the acceptability rate of patients to be recruited in a study proposing temperature monitoring at home, by a remote monitoring device or by the visit of an IDE at home (in association with the usual educational sessions), to children at risk of febrile neutropenia, from families with psycho-social vulnerabilities.

The main questions it aims to answer are:

* Will participants adhere to the telemonitoring system?
* Is the intervention feasible, in terms of the device's failure to record temperature data?
* Will parents behave appropriately when using the device?
* How satisfied will parents and caregivers be?
* What will be the physical tolerance of the device?
* On an exploratory basis, will the remote monitoring system be effective for months?

Researchers will compare :

* patients using the telemonitoring device for continuous temperature monitoring at home, in combination with education sessions on temperature monitoring and the device
* with patient with temperature monitoring at home by a nurse, 2 times a day, in combination with education sessions on temperature monitoring (without the telemonitoring device at home)

ELIGIBILITY:
Inclusion Criteria:

patient

* Aged 0 to 17 inclusive
* Followed in the Pediatric Onco-Hematology Department
* Primo-diagnosed with solid or hematological cancer (incident case)
* Having received a first cycle of chemotherapy
* Whose family has psycho-social vulnerabilities assessed by the Froger et al. tool, indicating a need for an IDE to support the family in monitoring the patient.

Exclusion Criteria:

Patient:

* with a dermatosis contraindicating the use of the device
* Refusing to participate in the study

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2028-05-04 (Estimated); Study Completion 2028-05-04 (Estimated)

PRIMARY OUTCOMES:
study acceptability rate | 24 months
  number of patients included/number of eligible patients offered the study.

IPD SHARING:
Plan to Share IPD: No